CLINICAL TRIAL: NCT05187832
Title: A Phase I Dose Escalation and Dose Expansion Study of AND019 in Patients With Estrogen Receptor Positive Human Epidermal Growth Factor Receptor 2 Negative Advanced or Metastatic Breast Cancer
Brief Title: A Study of AND019 in Women With ER Positive HER2 Negative Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AND019-MN-101
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AND019 single dose escalation and expansion (Experimental): Subjects will be administrated with AND019 capsule PO QD from 20 mg to 400 mg during Part 1, and 2 dose groups will be selected for dose expansion study
  Interventions: Drug: AND019 PO QD

INTERVENTIONS:
Drug: AND019 PO QD — AND019 administrated as oral capsule once per day for 28 days for each cycle

SUMMARY:
This is a first in human dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) activity, and preliminary anti-tumor activity of AND019 in postmenopausal women with advanced or metastatic estrogen receptor (ER)-positive (human epidermal growth factor receptor 2 [HER2]-negative) breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

1. Postmenopausal women defined as NCCN guideline at the time of informed consent.
2. Histological or cytological confirmation of advanced or metastatic ER+/HER2- breast cancer women who failed standard therapy or for which no standard therapy exists.
3. Prior therapy:

   1. No more than 1 line of chemotherapy for advanced breast cancer
   2. Recurrence or progression on at least one line of endocrine therapy in the advanced or metastatic disease setting and derived a clinical benefit from the endocrine therapy: Recurred or progressed while being treated with adjuvant endocrine therapy for a duration of at least 24 months, or progressed under endocrine therapy for more than 6 months in the advanced or metastatic setting
4. ECOG score 0-1.
5. Minimum life expectancy of a least 3 months as determined by the Investigator.
6. Evaluable disease per RECIST 1.1; for patients consent to tissue biopsy, disease suitable for tumor biopsy.
7. Sufficient bone marrow reserve and organ function.

Key Exclusion Criteria:

1. Previous treatment with any SERDs.
2. Patient any central nervous system metastasis.
3. Prior antitumor therapies:

   1. Received chemotherapies within 3 weeks before the first dose.
   2. Received systemic radiotherapy within 3 weeks before the first dose, or local radiotherapy within 7 days before the first dose
   3. Received other anti-tumor therapy such as endocrine therapy, immunotherapy, and target therapy within 3 weeks or 5 half-lives of the drug before the first dose of the study drug
   4. For bone metastasis, bisphosphonates and local remission therapy are allowed (7 days washout for local radiation therapy).
4. Patient who has participated in any other clinical trials for drugs or treatments within 5 half-lives for a prior investigational drug or 2 weeks from use of an investigational device prior to the first dose of study drug.
5. Patient who had major surgery or significant trauma within 4 weeks prior to the first dose of study drug (excluding needle biopsy), or has scheduled surgery during the study period.
6. Patient with serous unhealable wounds/ulcers/fractures within 4 weeks prior to the first dose of study drug.
7. Patient with adverse reactions to previous anti-tumor treatments who have not yet recovered to grade ≤1 according to CTCAE v5.0. (except for toxicities without safety risks as judged by Investigator, such as alopecia, grade 2 peripheral neuropathy etc.)
8. Patient who has used strong inhibitors or strong inducers of CYP3A, or grapefruit or grapefruit juice within 4 weeks prior to the first dose of study drug.
9. Patient unable to be administered oral medications or any condition that seriously affect digestion in the gastrointestinal tract at the judgement of the Investigator.
10. Patient with active infection within 1 week prior to the first dose of study drug, and currently need systemic anti-infective treatment.
11. Patient has a known history of the following: HIV infection without effective antiretroviral therapy (ART) or acceptable immune function, or syphilis infection, or HBsAg positive HBV or needs prophylaxis therapy or suppressive antiviral therapy before dosing, or has an HCV infection that hasn't completed curative antiviral treatment or with unacceptable viral load.
12. Patient has active cardiac disease or a history cardiac dysfunction.
13. Patient with third spacing that cannot be controlled clinically and is not suitable for the study by the Investigator's judgment.
14. Patient with known history of drug abuse.
15. Patient with mental disorder that, in the opinion of the Investigator, could lead to poor compliance with required study procedures.
16. Patient that cannot tolerate venous blood sampling.
17. Known to have other malignancy within the past 5 years, and is progressing or requires active treatment (except skin basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ who have received potentially radical treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events by severity, according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 | From baseline to 12 weeks after the last dose of study treatment (up to 25 months)
  Number of participants with adverse events
PK study of AND019 | At predefined timepoints at Day 1, Day 8, Day 15, and Day 22 of Cycle 1, and Day 1 of each cycle starting from Cycle 2 (each cycle is 28 days)
  Plasma concentration of AND019 over time

SECONDARY OUTCOMES:
Determine the RP2D | From baseline to up to the end of Cycle 1 (each cycle is 28 days)
  To observe the dose limiting toxicity (DLT) and maximum tolerated dose MTD to determine RP2D.
Percentage of Participants with Objective Response | Baseline and every 8 weeks from Cycle 1 Day 1 until Week 24, and then every 12 weeks until end of study treatment (up to 24 months) (each cycle is 28 days)
  ORR is defined as a complete response or partial response on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1)
Clinical Benefit Rate | Baseline and every 8 weeks from Cycle 1 Day 1 until Week 24 (each cycle is 28 days)
  CBR is defined as the percentage of participants achieving either of the following: confirmed complete response or partial response (as determined by the investigator according to RECIST v1.1); or the first occurrence of progressive disease after 24 weeks of study treatment.
Duration of Response | From the first occurrence of a documented objective response until first observation of disease progression or death from any cause on study, whichever occurs first (up to 24 months)
  DoR is defined as the percentage of participants achieving either of the following: confirmed complete response or partial response.

OTHER OUTCOMES:
Progression free survival | From treatment start date until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS is defined as the time from treatment start date until objective tumor progression (PD) or death whichever comes first
PD study of AND019 in blood samples | At predefined timepoints at baseline, Cycle 1 Day 15, Cycle 2 Day 1, and End of Treatment (up to 2 years) (each cycle is 28 days).
  Change from baseline in therapy resistant markers by liquid biopsy
PD study of AND019 in tissue samples | At predefined timepoints at baseline and between Cycle 2 Day 1 to Cycle 3 Day 28 (each cycle is 28 days)
  Change from baseline in therapy resistant markers by tissue biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD PhD, Study Director — Kind Pharmaceuticals LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States